CLINICAL TRIAL: NCT05742061
Title: Intra-articular Platelet Rich Plasma vs Corticosteroid in Treatment of Knee Osteoarthritis
Brief Title: Intra-articular Platelet Rich Plasma vs Corticosteroid in Treatment of Knee Osteoarthritis Patients
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Arwa El Sayed Abdel Rahman, Lecturer of Rheumatology, Rehabilitation and Physical Medicine, Benha University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MS 54-1-2023
Record Dates: First submitted 2023-02-01; First posted 2023-02-23 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Osteoarthritis Knee; Corticosteroid; Platelet Rich Plasma
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Adrenal Cortex Hormones

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- OA group injected by corticosteroid (Active Comparator): Group l include 50 patients who will be injected with one intra_articular injection of 2 ml of methylprednisolone acetate 40 mg/ml mixed with 2ml of lidocaine
  Interventions: Drug: Corticosteroid
- OA group injected by Platelet Rich Plasma (Active Comparator): Group lI include 50 patients who will be injected with a single 5 ml intra_articular injection of PRP prepared in our hospital
  Interventions: Other: Platelet Rich Plasma

INTERVENTIONS:
Drug: Corticosteroid — The injection will be given at a site near the superolateral pole of patella in the suprapatellar pouch under aseptic conditions and the patient will be advised to take one day of rest after injection and apply ice to the area if there are any signs of inflammation.
  Arms: OA group injected by corticosteroid
Other: Platelet Rich Plasma — PRP preparation :- 20 ml of venous blood will be drawn from the antecubital vein using an 18G needle to avoid traumatizing platelets and will be collected in a sterile tube containing 2 ml of Sodium Citrate anticoagulant. Approximately 2 ml of whole blood will be separated for a complete blood count.The blood with anticoagulant will centrifuged at 4000 rpm for 6-10 minutes to separate erythrocytes and then at 4000 rpm for 6-10 min to concentrate platelets.The final product was 4-5 ml of PRP containing leukocytes with platelet concentration of 3-5 times the average normal value.
  Arms: OA group injected by Platelet Rich Plasma

SUMMARY:
Knee osteoarthritis is the most common type of osteoarthritis in the lower extremity and constitutes 23% of all arthritis cases, about 13% of females and 10% of males aged above 60 years have symptomatic knee OA. Intra-articular corticosteroids (IACs) are a frequently-used treatment regimen for pain relief from symptomatic knee OA as it inhibits inflammation and reduces prostaglandin synthesis. Platelet-rich plasma (PRP) is an autologous blood product containing a high percentage of various growth factors (GFs), such as fibroblast growth factor, epidermal growth factor, vascular endothelial growth factor, transforming growth factor-β and platelet-derived growth factor. The aim of this study is to compare effect of intra-articular injection of platelet rich plasma versus corticosteroid in treatment of primary knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Patients 40-70 years of age suffering from knee OA with Kellgren Lawrence grade II or III on standing antero-posterior and lateral knee radiographs.
* Patients diagnosed according to ACR classification criteria.

Exclusion Criteria:

* Systemic diseases as Patients having diabetes mellitus,Cardiovascular diseases or coagulopathies.
* Those receiving treatment with anticoagulant , anti_platelet medications or systemic corticosteroid 10 days before injection or recent use of NSAIDs.
* Pregnant and breast feeding females.
* Patients have hemoglobin values <10 g/dl or platelet values<150,000/ml.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Patients 40-70 years of age suffering from knee OA
Enrollment: 100 (Estimated)
Dates: Start 2023-04 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Assessment of knee pain, stiffness and physical function prior knee injection | Assessment will be done just before injection
  Assessment through the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) score. The final score for the WOMAC was determined by adding the aggregate scores for pain, stiffness, and function. Scores range from 0 to 96 for the total WOMAC where 0 represents the best health status and 96 the worst possible status.
Assessment of knee pain, stiffness and physical function 2 weeks after injection | 2 weeks after injection
  Assessment through WOMAC score
Assessment of knee pain, stiffness and physical function 6 weeks after injection | 6 weeks after injection
  Assessment through WOMAC score
Assessment of knee pain, stiffness and physical function 12 weeks after injection | 12 weeks after injection
  Assessment through WOMAC score

IPD SHARING:
Plan to Share IPD: No